CLINICAL TRIAL: NCT04360577
Title: Effect of Acupuncture for Quality of Life and Symptom Control in Patients With Gastric Cancer Undergoing Adjuvant Chemotherapy
Brief Title: Acupuncture for QoL and Symptoms in Gastric Cancer During Adjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Hospital of Nanjing University of Traditional Chinese Medicine (Unknown); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Southern Medical University, China (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); First People's Hospital of Foshan (Other); Yuebei People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018KT1226-2; 2017YFC1700603 (Other Grant/Funding Number: The National Key Research and Development Program of China)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Stomach Neoplasms
Keywords: Gastric Cancer; Acupuncture; Quality of Life; Symptom Burden; Adjuvant Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose acupuncture (Experimental): Acupuncture for 7 times every 3 weeks (one cycle of chemotherapy) for 9 weeks (3 cycles of chemotherapy)
  Interventions: Procedure: acupuncture
- Low-dose acupuncture (Experimental): Acupuncture for 3 times every 3 weeks (one cycle of chemotherapy) for 9 weeks (3 cycles of chemotherapy)
  Interventions: Procedure: acupuncture
- Usual care (No Intervention): Chemotherapy without acupuncture

INTERVENTIONS:
Procedure: acupuncture — Acupuncture at back-shu points according to heat-pain threshold measurement at 24 well-points, combing with electro-acupuncture at Baihui(GV20), Yintang(GV29), Neiguan(PC6), Zusanli(ST36), and Gongsun(SP4).
  Arms: High-dose acupuncture; Low-dose acupuncture

SUMMARY:
In the investigator's pilot study(NCT 03753399), a trend of improvement of quality of life, as well as release of symptoms, in gastric patients in acupuncture groups was indicated. This study will evaluate the efficacy of acupuncture on QoL in gastric cancer patients undergoing postoperative adjuvant chemotherapy with more samples. Enrolled participates will randomly receive high-dose acupuncture, low-dose acupuncture or non-acupuncture during the first 3 cycles of adjuvant chemotherapy after resection.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pathologically diagnosed with gastric cancer or esophagogastric junction cancer after R0 resection and D2 lymph node dissection;
* 2.Pathological stage II or stage III
* 3.Without tumor recurrence confirmed by image examination;
* 4.No chemotherapy after surgery, planning to accept at least 3 cycles of adjuvant chemotherapy;
* 5.Age:18~75 years old
* 6.ECOG score≤ 2
* 7. Normal organ function, including: 7.1 Bone marrow function: absolute neutrophil count (ANC)≥1.5×10e9/L, platelet (PLT)≥100×10e9/ L,hemoglobin (Hb)≥90g/L; 7.2 Kidney function: Serum creatinine (Scr)≤1.5mg/dl(133μmol/L), or creatinine clearance rate (Ccr)≥60ml/min; 7.3 Liver function: Total bilirubin (TB)≤1.5×upper limit of normal value (ULN), Alanine transaminase (ALT)≤2.5×ULN, Aspartate transaminase (AST)≤2.5×ULN;
* 8. Can understand the study well and finish the questionnaires in this study; 9. With the written informed consent.

Exclusion Criteria:

* 1. Can not finish the baseline assessment;
* 2. Needle phobia;
* 3. Currently diagnosed with psychiatric disorder (e.g., severe depression, obsessive-compulsive disorder, or schizophrenia);
* 4. History of autoimmune diseases, hematological diseases or organ transplantation, or long term use of hormones or immunosuppressors;
* 5. Implanted with heart pacemaker;
* 6. Has accepted neoadjuvant radiotherapy before surgery;
* 7. Planning to accept adjuvant radiotherapy after surgery;
* 8. With active infection;
* 9. Acupuncture treatment within the previous 6 weeks;
* 10.Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Total AUC of FACT-Gastric TOI | At the end of Cycle 3 ( 21 days for one cycle)
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. FACT-Gastric TOI is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS) of the FACT-Gastric Scoring. The range of FACT-Gastric TOI is 0-132. The higher the score, the better the quality of life. TOI for each patient will be recorded at baseline and once a week during the 3 cycles of chemotherapy (21 days for one cycle). The area under curve (AUCs) for each week are calculated by linear interpolation respectively, and then added together for the total AUC during the 3 cycles of chemotherapy.

SECONDARY OUTCOMES:
Average trajectory of FACT-Gastric TOI over time | Baseline(at randomization), once a week during the 3 cycles of treatment (21 days for 1 cycle)
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. FACT-Gastric TOI is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS) of the FACT-Gastric Scoring. The range of FACT-Gastric TOI is 0-132. The higher the score, the better the quality of life.
Total AUC of FACT-Gastric Scoring | At the end of Cycle 3 ( 21 days for one cycle)
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. It is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, SOCIAL WELL BEING (SWB) SUBSCALE, EMOTIONAL WELL BEING (EWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS). The range of FACT-Gastric scoring is 0-184. The higher the score, the better the quality of life. FACT-Gastric scoring for each patient will be recorded at baseline and once a week during the 3 cycles of chemotherapy (21 days for one cycle). The area under curve (AUCs) for each week are calculated by linear interpolation respectively, and then added together for the total AUC during the 3 cycles of chemotherapy.
Average trajectory of FACT-Gastric Scoring over time | Baseline(at randomization), once a week during the 3 cycles of treatment (21 days for 1 cycle)
  FACT-Gastric Scoring is designed for measurement of quality of life(QoL) for gastric cancer patients. It is composed of PHYSICAL WELL BEING (PWB) SUBSCALE, SOCIAL WELL BEING (SWB) SUBSCALE, EMOTIONAL WELL BEING (EWB) SUBSCALE, FUNCTIONAL WELL BEING (FWB) SUBSCALE, and GASTRIC CANCER SUBSCAL (GaCS). The range of FACT-Gastric scoring is 0-184. The higher the score, the better the quality of life.
Total AUC of GASTRIC CANCER SUBSCAL (GaCS) of FACT-Gastric | At the end of Cycle 3 ( 21 days for one cycle)
  The GaCS of FACT-Gastric focuses on the symptoms and functions related to gastric cancer specifically. The range of GaCS is 0-76. The higher the score, the better the quality of life. GaCS for each patient will be recorded at baseline and once a week during the 3 cycles of chemotherapy (21 days for one cycle). The area under curve (AUCs) for each week are calculated by linear interpolation respectively, and then added together for the total AUC during the 3 cycles of chemotherapy.
Average trajectory of GASTRIC CANCER SUBSCAL (GaCS) of FACT-Gastric | Baseline(at randomization), once a week during the 3 cycles of treatment (21 days for 1 cycle)
  The GaCS of FACT-Gastric focuses on the symptoms and functions related to gastric cancer specifically. The range of GaCS is 0-76. The higher the score, the better the quality of life.
Total AUC of Modified Edmonton Symptom Assessment Scale | At the end of Cycle 3 ( 21 days for one cycle)
  Edmonton symptom assessment scale (ESAS) is a questionnaire used for symptom assessment in cancer patients. It was composed of 10 items with score range of 0-10 for each item, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, shortness of breath, and other. ESAS was then modified in 2015, with additional symptoms of constipation and sleep. The higher the score, the worse the symptom is. ESAS scoring for each patient will be recorded everyday in the first week, and then once a week in the next 2 weeks during each cycle of chemotherapy (21 days for 1 cycle). The AUCs are calculated by linear interpolation respectively, and then added together for the total AUC during the 3 cycles of chemotherapy.
Average trajectory of Modified Edmonton Symptom Assessment Scale | Everyday in the first week, then once a week in the next 2 weeks during each cycle of chemotherapy (21 days for 1 cycle)
  Edmonton symptom assessment scale (ESAS) is a questionnaire used for symptom assessment in cancer patients. It was composed of 10 items with score range of 0-10 for each item, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing, shortness of breath, and other. ESAS was then modified in 2015, with additional symptoms of constipation and sleep. The higher the score, the worse the symptom is.

OTHER OUTCOMES:
Concentration of circulating myeloid-derived suppressor cells | At the end of Cycle 3 ( 21 days for one cycle)
  Myeloid-derived suppressor cells in peripheral blood will be detected using flow cytometry
Concentration of circulating Treg cells | At the end of Cycle 3 ( 21 days for one cycle)
  Treg cells in peripheral blood will be detected using flow cytometry
Number of Circulating tumor cells | At the end of Cycle 3 ( 21 days for one cycle)
  Circulating tumor cells in peripheral blood will be detected using microfluidic chip
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Adverse events will be assessed during the period of 3 cycles of treatment (21 days for each cycle), since the date of randomization. Adverse events will be recorded once any side effect happens.
  Treatment-emergent adverse events is defined as any adverse events happened after randomization. The severity is validated using NCI-CTCAE V4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Prof., Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (11):
- China (11):
  - Foshan First People's Hospital, Foshan, Guangdong
  - The first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sixth affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The first affiliated hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Fifth affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - Affiliated Hospital of Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
IPD can be obtained from the PI with application after article publication.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Zhu YJ, Chang XS, Wu XY, Wang W, Diao DC, Li Y, Zhang HY, Xiao J, Zhai XH, Yu JL, Wang W, Zhou JX, Huang ZL, Zhang T, Ouyang W, Janjigian YY, Cytryn SL, Xiao ZZ, Liu YH, Zhou R, Ma HC, Chen YD, Peng JJ, Mao JJ, Zhang HB. Electro-acupuncture for quality of life during adjuvant chemotherapy in gastric cancer: a randomized trial. J Natl Cancer Inst. 2025 Oct 27:djaf309. doi: 10.1093/jnci/djaf309. Online ahead of print. PMID 41143548
- [Derived] Chang X, Zhu Y, Zhao W, Liu Y, He Y, Chen Y, Xu D, Mao JJ, Zhang HB. Electro-acupuncture for health-related quality of life and symptoms in patients with gastric cancer undergoing adjuvant chemotherapy (EAGER): a protocol for a multicenter randomized controlled trial. Health Qual Life Outcomes. 2023 Jul 11;21(1):70. doi: 10.1186/s12955-023-02135-9. PMID 37434165